CLINICAL TRIAL: NCT00462748
Title: A MC, DB, Rand, Study to Evaluate Efficacy, Safety and Tolerability of Eze/Simva 10/40 mg, Atorva 40 mg, Rosuva 10 mg in Achieving LDL-C <2 mmol/l in Pts With CVD...on Simva 40 mg With LDL-C ³2 mmol/l
Brief Title: A Study to Determine the Number of Patients Who Reach Optimal Cholesterol Levels on Each of Three Different Treatments (0653A-121)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0653A-121; MK0653A-121; 2007_013
Record Dates: First submitted 2007-04-18; First posted 2007-04-19 (Estimated); Results first posted 2009-08-17 (Estimated); Last update posted 2024-05-16 (Actual); Status verified 2022-02

CONDITIONS: Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia | interventions — Ezetimibe, Simvastatin Drug Combination; Atorvastatin; Rosuvastatin Calcium

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- 1 (Experimental): Arm 1: Drug
  Interventions: Drug: ezetimibe (+) simvastatin
- 2 (Active Comparator): Arm 2: Active comparator
  Interventions: Drug: Comparator: atorvastatin
- 3 (Active Comparator): Arm 3: Active comparator
  Interventions: Drug: Comparator: rosuvastatin

INTERVENTIONS:
Drug: ezetimibe (+) simvastatin — ezetimibe (+) simvastatin 10/40mg. once daily tablet formulation, all tablet form, taken orally, cholesterol lowering medication.
  Other Names: MK0653A
  Arms: 1
Drug: Comparator: atorvastatin — atorvastatin 40mg. once daily tablet formulation, all tablet form, taken orally
  Other Names: atorvastatin
  Arms: 2
Drug: Comparator: rosuvastatin — rosuvastatin 10 mg. once daily tablet formulation, all tablet form, taken orally.
  Other Names: rosuvastatin
  Arms: 3

SUMMARY:
To evaluate the percentage of patients with either established cardiovascular disease (CVD), at "high risk" of developing CVD or with diabetes who are on simvastatin 40mg, with fasting LDL-C > 2mmol/l, who are able to attain the recommended LDL-C target of < 2mmol/l following 6 weeks treatment with either ezetimibe/simvastatin 10/40mg, atorvastatin 40mg or rosuvastatin 10mg.

ELIGIBILITY:
Inclusion Criteria:

* Patient Is Male Or Female And Aged Over 18
* Patient Provides Written Informed Consent
* Patient Has A Fasting Ldl-C Level >2mmol/L At Both Visit 1 And Again At Visit 2
* Patient Has Established Cvd, Diabetes Or At "High Risk" Of Cvd (>20 % Risk Over 10 Years, Framingham Scale)
* Patient Has Taken Simvastatin 40mg Continuously For The Past 6 Weeks
* Patient Has A Fasting Triglyceride Level Of <3.7mmol/L
* Patient Has Hba1c <9% At Visit 1
* Patient Is 75% Compliant With Medication Between Visit 1 And Visit 2

Exclusion Criteria:

* Patient Is Hypersensitive To Any Of The Study Medications Or Their Components
* Patient Has A History Of, Or Active Liver Disease (Persistent Elevation Of Alt / Ast (>3xuln)
* Patient Is Pregnant, Lactating, Or A Female Patient Of Childbearing Potential Not Using Adequate Contraception
* Patient Has Severe Renal Impairment: Creatinine Clearance <30ml/Min (Cockcroft-Gault Equation) (In Patients With Moderate Renal Impairment: <60ml/Min, The Dose Of Rosuvastatin Will Be 5mg In Line With The Spc)
* Patient Has Uncontrolled Endocrine Or Metabolic Disease Known To Influence Serum Lipids Or Lipoproteins (I.E. Secondary Causes Of Hyperlipidaemia Such As Hypothyroidism Or Hyperthyroidism)
* Patient Has A Recent History Of, Or Current, Alcohol Abuse
* Patient Has Ck >10 X Uln At Visit 1 Or Visit 2
* Patient Has Fasting Ldl-C >4.2mmol/L
* Patient Has Any Acute Or Serious Condition, Or History Suggestive Of Myopathy Or Predisposing To The Development Of Renal Failure Secondary To Rhabdomyolysis (E.G. Sepsis, Hypotension, Major Surgery, Trauma, Severe Metabolic, Severe Endocrine And Electrolyte Disorders Or Uncontrolled Seizures)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 786 (Actual)
Dates: Start 2007-03; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] McCormack T, Harvey P, Gaunt R, Allgar V, Chipperfield R, Robinson P; IN-PRACTICE study. Incremental cholesterol reduction with ezetimibe/simvastatin, atorvastatin and rosuvastatin in UK General Practice (IN-PRACTICE): randomised controlled trial of achievement of Joint British Societies (JBS-2) cholesterol targets. Int J Clin Pract. 2010 Jul;64(8):1052-61. doi: 10.1111/j.1742-1241.2010.02429.x. Epub 2010 May 12. PMID 20487050

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients with diabetes, cardiovascular disease (CVD) or a "high risk" of developing CVD and a fasting LDL-C level of ≥2mmol/l, having been on simvastatin 40mg for 6 weeks were assigned to 10/40 mg ezetimibe/simvastatin; 40 mg atorvastatin; 10 mg rosuvastatin (5 mg in elderly/Asian patients (in line with UK SPC)) between 27/03/2007 and 31/03/2008
Pre-assignment Details: All patients were subjected to a 6 week run-in period on open label 40 mg simvastatin to stabilise their LDL-C levels. Patients whose LDL-C at the end of this period was below 2.0 mmol/l or who were <75% compliant with run-in medication, were excluded from the study
Groups:
- Ezetimibe/Simvastatin: ezetimibe (+) simvastatin 10/40mg. once daily tablet formulation, all tablet form, taken orally
- Atorvostatin: atorvastatin 40mg. once daily tablet formulation, all tablet form, taken orally
- Rosuvastatin: rosuvastatin 10 mg. once daily tablet formulation, all tablet form, taken orally
Period: Overall Study
Arm/Group | Ezetimibe/Simvastatin | Atorvostatin | Rosuvastatin
Started | 261 | 263 | 262
Completed | 249 | 252 | 251
Not Completed | 12 | 11 | 11
Not completed — Adverse Event | 7 | 5 | 9
Not completed — Protocol Violation | 0 | 2 | 1
Not completed — Withdrew consent | 3 | 3 | 0
Not completed — Lost to Follow-up | 1 | 1 | 1
Not completed — Discontinued after 41 days Rx | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ezetimibe/Simvastatin | Atorvostatin | Rosuvastatin | Total
Number analyzed (Participants) | 261 | 263 | 262 | 786
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.7 (8.65) | 64.2 (8.44) | 63.9 (8.61) | 64.3 (8.56)
Age, Customized [Number; unit: participants]
  < 70 years | 185 | 187 | 195 | 567
  >=70 years | 76 | 76 | 67 | 219
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 101 | 78 | 84 | 263
  Male | 160 | 185 | 178 | 523
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian | 3 | 0 | 2 | 5
  White | 254 | 261 | 257 | 772
  Black | 4 | 0 | 2 | 6
  Other | 0 | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients Achieving a Target of Fasting LDL-C of <2mmol/l at Study End
Description: Fasting LDL-C was the primary efficacy variable. The primary efficacy analysis was based on the proportion of patients achieving a target of <2mmol/l in fasting LDL-C at study end.
Time Frame: 6 Weeks
Population: The Full Analysis Set (FAS) all patients who were:
  * Randomised
  * Took at least one dose of double-blind medication
  * Had a baseline measurement of efficacy
  * Had a post-baseline measurement of efficacy
  Patients were analysed according to the treatment group they were randomised, regardless of the treatment they received
Measure: Number; unit: Percent
Arm/Group | Ezetimibe/Simvastatin | Atorvostatin | Rosuvastatin
Number analyzed (Participants) | 255 | 259 | 258
Percent | 67.4 | 36.3 | 17.4
Statistical Analysis 1: Comparison: Ezetimibe/Simvastatin vs Atorvostatin; Ho is no difference in proportion achieving the target of LDL-C < 2mmol/l.. 240 patients per group give a power of at least 85% to detect a 15% difference in this proportion, assuming the percentage decrease from baseline in LDL-C was 25% in the E/S group and 15% in the two comparator groups. A two-sided 0.025 test to allow for multiple comparisons was used; Test type: Superiority or Other; p < 0.001, Regression, Logistic — Hochberg's FDR was used to power the study; the power was based on a two-sided p value of 0.025; The logistic regression model included terms for treatment and stratum; treatment by stratum interaction was assessed
Statistical Analysis 2: Comparison: Ezetimibe/Simvastatin vs Rosuvastatin; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, Regression, Logistic — Hochberg's FDR was used to power the study; the power was based on a two-sided p value of 0.025; The logistic regression model included terms for treatment and stratum; treatment by stratum interaction was assessed

ADVERSE EVENTS:
Arm/Group | Ezetimibe/Simvastatin | Atorvostatin | Rosuvastatin
Serious Adverse Events (participants affected / at risk) | 4 | 2 | 4
Other Adverse Events (participants affected / at risk) | 6 | 1 | 8
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk (number of events):
Term (organ system) | Ezetimibe/Simvastatin | Atorvostatin | Rosuvastatin
Platelet count decreased (Investigations) | 1/259 (1) | 0/260 (0) | 0/261 (0)
Aortic regurgitation (Cardiac disorders) | 1/259 (1) | 0/260 (0) | 0/261 (0)
Chest pain (General disorders) | 1/259 (1) | 0/260 (0) | 0/261 (0)
Oesophageal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/259 (1) | 0/260 (0) | 0/261 (0)
Erthematous rash (Skin and subcutaneous tissue disorders) | 0/259 (0) | 1/260 (1) | 0/261 (0)
Areterial haemorrhage (Vascular disorders) | 0/259 (0) | 1/260 (1) | 0/261 (0)
Rectal bleeding (Gastrointestinal disorders) | 0/259 (0) | 0/260 (0) | 1/261 (1)
Hydronephrosis (Renal and urinary disorders) | 0/259 (0) | 0/260 (0) | 1/261 (1)
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/259 (0) | 0/260 (0) | 1/261 (1)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0/259 (0) | 0/260 (0) | 1/261 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected / at risk (number of events):
Term (organ system) | Ezetimibe/Simvastatin | Atorvostatin | Rosuvastatin
Diarrhea (Gastrointestinal disorders) | 6/259 (6) | 1/260 (1) | 8/261 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.